CLINICAL TRIAL: NCT05716035
Title: A Phase III, Open-label Extension Trial of tMG to Evaluate the Safety and Efficacy of Tocilizumab in Subjects With Generalized Myasthenia Gravis (gMG)
Brief Title: Open-Label Extension of Tocilizumab in Subjects With Generalized Myasthenia Gravis
Acronym: tMG-E
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tang-Du Hospital (Other)
Responsible Party: Principal Investigator, changting, Associate Professor, Tang-Du Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: V1.0, 20221201
Record Dates: First submitted 2023-01-27; First posted 2023-02-08 (Actual); Last update posted 2024-01-22 (Actual); Status verified 2024-01

CONDITIONS: Myasthenia Gravis, Generalized
Keywords: Generalized Myasthenia Gravis; Tocilizumab; Open-label
MeSH Terms: conditions — Myasthenia Gravis | interventions — tocilizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- tocilizumab (Experimental): Participants will receive tocilizumab 8mg/Kg administered intravenously (IV) on weeks 1,5,9 and 13 of the open-lable period.
  Interventions: Drug: Tocilizumab Injection

INTERVENTIONS:
Drug: Tocilizumab Injection — Participants will receive IV tocilizumab

SUMMARY:
To evaluate the safety and efficacy of tocilizumab in the treatment of generalized myasthenia gravis (gMG) as an extension study for the participants who previously completed Study tMG(NCT05067348).

DETAILED DESCRIPTION:
tMG-E was an extension study designed to provide the participants who completed Study tMG an opportunity to receive tocilizumab and collect clinical data to provide long-term safety and efficacy information on tocilizumab in participants with gMG.

After receiving blinded study treatment (tocilizumab or placebo) in Study tMG for 16 weeks, participants were eligible to enroll in the tMG-E extension study. Participants were to enter Study tMG-E within 8 weeks after completing their Week 16 visit in Study tMG.

Study tMG-E consisted of an Open-Label treatment Phase up to 16 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Participant has completed Study tMG.
2. Participant has given written informed consent.
3. MG-ADL score ≥ 5 points, or a decrease of ≤ 3 points relative to the baseline MG-ADL of the tMG study

Exclusion Criteria:

1. Participants had clinically relevant active infections (such as sepsis, pneumonia, or abscess) or severe infections (resulting in hospitalization or requiring antibiotic treatment) in the past 4 weeks;
2. Those with high-risk tuberculosis infection, acquired tuberculosis infection, and chronic hepatitis after the tMG study;
3. planned thymectomy during RCP;
4. Received IVIG or plasma exchange in the past 4 weeks;
5. Any medical condition or circumstances that, in the opinion of the investigator, might have interfered with the participant's participation in the study, posed any added risk for the participant, or confounded the assessment of the participants.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2023-04-01 (Actual); Primary Completion 2024-07-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of treatment-emergent adverse events (TEAEs) | From Baseline (Day 1) to Safety Follow-Up Visit (up to 16 weeks)

SECONDARY OUTCOMES:
Change in Quantitative Myasthenia Gravis (QMG) scores. | 16 weeks
Proportion of subjects with both (1) ≥ 3-point improvement in QMG and (2) lasts ≥4 weeks | 16 weeks
Proportion of subjects with both (1) ≥ 2-point improvement in MG-ADL and (2) lasts ≥4 weeks | 16 weeks
Change from baseline in Myasthenia Gravis Activities of Daily Living (MG-ADL) Profile score | 16 weeks
Change in Myasthenia Gravis Composite (MGC) score | 16 weeks
Change in Myasthenia Gravis Quality of Life-15, revised (MG-QOL15r) score. | 16 weeks

CONTACTS AND LOCATIONS:
Locations (6):
- China (6):
  - Beijing Tiantan Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Xiangya Hospital Central South University, Changsha, Hunan
  - Tangdu Hospital, The Fourth Military Medical University, Xi'an, Shaanxi
  - Huashan Hospital, Shanghai, Shanghai Municipality
  - West China Hospital of Sichuan University, Chengdu, Sichuan
  - Tianjin medical university general hospital, Tianjin, Tianjin Municipality

IPD SHARING:
Plan to Share IPD: No